CLINICAL TRIAL: NCT01322711
Title: Effects on Oxidative Stress, Coagulation, Platelet Activation and Inflammatory Indexes of Atorvastatin and/or Aspirin Treatment in Patients at High Risk of Vascular Events
Brief Title: Atorvastatin, Aspirin, Oxidative Stress, Coagulation and Platelet Activation Indexes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Stefania Basili, Prof., University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATORVASA
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus; Hypercholesterolemia
Keywords: Thromboxane; Aspirin; Atorvastatin; Platelet activation; Thrombin Activation; Oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): Each day accordingly to randomization patients allocated to Atorvastatin received a pill of 40 mg of atorvastatin. In diabetic patients the concomitant aspirin treatment include a previous 30 days treatment with 100 mg daily of aspirin.
  All patients followed the diet used in the placebo group.
  Interventions: Drug: Atorvastatin
- Diet (Placebo Comparator): Low-fat diet with mean macronutrient profiles that were close to the present Adult Treatment Panel III guidelines (7% energy from saturated fat and, 200 mg dietary cholesterol per day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40 mg day
  Other Names: Totalip 40 mg; Torvast 40 mg
  Arms: Atorvastatin
Drug: Placebo — Diet
  Arms: Diet

SUMMARY:
Primary and secondary prevention trials with statins, as well as with antiplatelet, clearly demonstrated that these drugs are able to reduce cardiovascular events. Even if the principal mechanism of action of statins is to lower cholesterol, other effects, the so-called pleiotropic effects, have been considered as adjunctive properties potentially accounting for the anti-atherosclerotic effect of statins.

Inhibition of oxidative stress may be considered an intriguing pleiotropic effect in view of the fact that oxidative stress is thought to be a key event in the initiation and progression of atherosclerotic disease. Reduction of several markers of oxidative stress including isoprostanes, 8-hydroxydeoxyguanosine (8-OHdG), and nitrotyrosine have been observed after statin treatment. NADPH oxidase is among the most important sources of reactive oxygen species involved in atherosclerotic disease. The investigators developed an ELISA to evaluate serum levels of soluble-gp91phox, the catalytic core of phagocyte NADPH oxidase. Recently the investigators showed that statins (30 days treatment) exert an antioxidant effect via inhibition of soluble gp91phox expression.

The exact mechanism by which atorvastatin reduces NADPH oxidase, however, is unclear. Recent study showed that statin treatment inhibits leukocyte ROCK activity, a protein kinase implicated in the activation of NADPH oxidase, with a mechanism that seems to be independent from lowering cholesterol. To further study the mechanism(s) implicate in gp91phox downregulation by statin the investigators planned the present study in patients with high risk of vascular events such as hypercholesterolemic and Type 2 Diabetes mellitus patients.

In addition the investigators want to evaluate the synergistic role of atorvastatin with aspirin treatment.

DETAILED DESCRIPTION:
Primary and secondary prevention trials with statins, as well as with antiplatelet, clearly demonstrated that these drugs are able to reduce cardiovascular events. Even if the principal mechanism of action of statins is to lower cholesterol, other effects, the so-called pleiotropic effects, have been considered as adjunctive properties potentially accounting for the antiatherosclerotic effect of statins.

Inhibition of oxidative stress may be considered an intriguing pleiotropic effect in view of the fact that oxidative stress is thought to be a key event in the initiation and progression of atherosclerotic disease. Reduction of several markers of oxidative stress including isoprostanes, 8-hydroxydeoxyguanosine (8-OHdG), and nitrotyrosine have been observed after statin treatment. NADPH oxidase is among the most important sources of reactive oxygen species involved in atherosclerotic disease. The investigators developed an ELISA to evaluate serum levels of soluble-gp91phox, the catalytic core of phagocyte NADPH oxidase. Recently the investigators showed that statins (30 days treatment) exert an antioxidant effect via inhibition of soluble gp91phox expression.

The exact mechanism by which atorvastatin reduces NADPH oxidase, however, is unclear. Recent study showed that statin treatment inhibits leukocyte ROCK activity, a protein kinase implicated in the activation of NADPH oxidase, with a mechanism that seems to be independent from lowering cholesterol.

Accelerated atherosclerosis is a typical feature of type 2 diabetes mellitus (T2DM). Thus, patients with T2DM have a 2- to 4-fold increased risk of cardiovascular diseases (CAD) and 2- to 6-fold increased risk of stroke.

Platelets play a major role in the etiology of atherosclerotic disease, as shown by the significant decrease of cardiovascular events in patients treated with aspirin, an inhibitor of COX1 that prevents platelet thromboxane (Tx) A2 formation. Despite this, interventional trials with aspirin in diabetic patients failed to show a beneficial effect. It has been previously demonstrated that COX1 inhibition determines a shift in arachidonic acid metabolism towards other pathways, such as the lipooxygenase system. The investigators speculate that COX1 inhibition could also be associated with increased conversion of arachidonic acid to platelet isoprostane formation; the increase of platelet isoprostanes would balance the inhibition of TxA2, thus hampering the antiplatelet effect of aspirin. As reported above, statins have been reported to down-regulate systemic isoprostanes with a mechanism that may involve inhibition of NADPH oxidase,therefore it could be interesting to examine if statins improve the antiplatelet effect of aspirin via inhibition of platelet isoprostanes.

To further study the mechanism(s) implicate in gp91phox downregulation by statin the investigators planned the present study in patients with hypercholesterolemia.

Furthermore, the second part of the study will be addressed to evaluate the synergistic role of atorvastatin with aspirin treatment in Type 2 Diabetes mellitus patients.

ELIGIBILITY:
For Hypercholesterolemic patients:

Inclusion Criteria:

* Patients with polygenic hypercholesterolemia (LDL-C > 160 mg/dl)
* Males and Females
* White race
* Sign of the informed consent

Exclusion Criteria:

* Liver insufficiency
* Serious renal disorders
* Diabetes mellitus
* Arterial hypertension
* History or evidence of previous myocardial infarction or other atherothrombotic diseases
* Any autoimmune diseases
* Cancer
* Present or recent infections
* Patients were taking nonsteroidal antiinflammatory drugs, drugs interfering with cholesterol metabolism, or vitamin supplements

For T2 Diabetic patients:

Inclusion Criteria:

* Patients with T2DM diagnosed according to the American Diabetes Association definition
* Treatment with 100 mg/day aspirin from at least 30 days
* Males and Females
* White race
* Sign of the informed consent

Exclusion Criteria:

* recent history (< 3 months) of acute vascular events
* clinical diagnosis of type 1 DM
* serum creatinine level greater than 2.5 mg/dl
* active infection or malignancy
* cardiac arrhythmia or congestive heart failure
* use of non-steroidal anti-inflammatory drugs, vitamin supplements, or other antiplatelet drugs such as clopidogrel in the previous 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of effect of Atorvastatin Therapy in Hypercholesterolemic Patients (n=30) and Diabetic Patients (n=30) | Baseline, 2 hours, 24 hours, 3 days, 7 days, 30 days
  In Hypercholesterolemic patients (n=30) and in Diabetic patients (n=30) under chronic treatment with low dose aspirin (100 mg daily for at least 30 days), blood and urine samples were taken at each above reported time to evaluate the effect of atorvastatin or no treatment (Diet) on platelet recruitment, platelet and serum isoprostanes, platelet and serum thromboxane A2, platelet and serum NOX2 activation indexes, thrombin activation indexes, urinary excretion of thromboxane and isoprostanes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Basili, Prof., Principal Investigator — Sapienza-Univerity of Rome
Locations (1):
- Stefania Basili, Rome, Italy

REFERENCES:
- [Background] Carnevale R, Pignatelli P, Di Santo S, Bartimoccia S, Sanguigni V, Napoleone L, Tanzilli G, Basili S, Violi F. Atorvastatin inhibits oxidative stress via adiponectin-mediated NADPH oxidase down-regulation in hypercholesterolemic patients. Atherosclerosis. 2010 Nov;213(1):225-34. doi: 10.1016/j.atherosclerosis.2010.08.056. Epub 2010 Aug 19. PMID 20832062
- [Background] Pignatelli P, Carnevale R, Cangemi R, Loffredo L, Sanguigni V, Stefanutti C, Basili S, Violi F. Atorvastatin inhibits gp91phox circulating levels in patients with hypercholesterolemia. Arterioscler Thromb Vasc Biol. 2010 Feb;30(2):360-7. doi: 10.1161/ATVBAHA.109.198622. Epub 2009 Dec 3. PMID 19965781
- [Derived] Pignatelli P, Carnevale R, Pastori D, Cangemi R, Napoleone L, Bartimoccia S, Nocella C, Basili S, Violi F. Immediate antioxidant and antiplatelet effect of atorvastatin via inhibition of Nox2. Circulation. 2012 Jul 3;126(1):92-103. doi: 10.1161/CIRCULATIONAHA.112.095554. Epub 2012 May 21. PMID 22615342